CLINICAL TRIAL: NCT00284154
Title: A Phase II Trial of VInflunine in the Treatment of Patients With Relapsed Extensive Small Cell Lung Cancer
Brief Title: Vinflunine in the Treatment of Patients With Relapsed Extensive Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LUN 122
Record Dates: First submitted 2006-01-27; First posted 2006-01-31 (Estimated); Results first posted 2013-03-13 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-02

CONDITIONS: Carcinoma, Small Cell; Lung Cancer
Keywords: Extensive stage; Relapsed
MeSH Terms: conditions — Carcinoma, Small Cell; Lung Neoplasms; Recurrence | interventions — vinflunine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Patients received vinflunine 320 mg/m2 every 21 days as a 15- to 20-minute infusion.
  Interventions: Drug: Vinflunine

INTERVENTIONS:
Drug: Vinflunine — 320mg/m2 every 21 days as a 15-20 minute infusion
  Other Names: Javlor

SUMMARY:
This clinical trial involves the administration of the chemotherapeutic medication vinflunine. Vinflunine is not approved by the FDA and is experimental in the treatment of extensive small cell lung cancer. The purpose of this research trial is to study the effectiveness of vinflunine in patients with relapsed extensive small cell lung cancer, evaluate the toxicity, and evaluate how long the response to this drug lasts.

DETAILED DESCRIPTION:
Eligible patients will receive vinflunine as a 15-20 minute intravenous (IV)infusion once every three weeks (21 days). This three week treatment period is called a cycle. Patients whose cancer has not grown or if it has decreased in size may receive up to 6 cycles of vinflunine. Evaluation will be conducted every other cycle.

ELIGIBILITY:
Inclusion Criteria:

* Small cell lung cancer with progression after one previous chemotherapy or chemotherapy/radiation therapy regimen
* Measurable or evaluable disease
* Able to perform activities of daily living with minimal assistance
* Adequate hematological, liver, and kidney function
* Must give written informed consent prior to entry

Exclusion Criteria:

* CNS involvement
* Serious active infection or underlying medical condition
* Significant history of uncontrolled cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2006-01; Primary Completion 2009-05 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R. Spigel, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (3):
- United States (3):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Oncology Hematology Care, Cincinnati, Ohio
  - Tennessee Oncology, PLLC, Nashville, Tennessee

REFERENCES:
- [Result] Spigel DR, Hainsworth JD, Lane CM, Clark B, Burris HA, Greco FA. Phase II trial of vinflunine in relapsed small cell lung cancer. J Thorac Oncol. 2010 Jun;5(6):874-8. doi: 10.1097/jto.0b013e3181d86b76. PMID 20521355
- See also: Published article in the Journal of Thoracic Oncology — http://journals.lww.com/jto/pages/articleviewer.aspx?year=2010&issue=06000&article=00020&type=abstract

RESULTS

PARTICIPANT FLOW:
Groups:
- Vinflunine: Patients received vinflunine 320 mg/m2 every 21 days as a 15- to 20-minute infusion.
Period: Overall Study
Arm/Group | Vinflunine
Started | 51
Completed | 9
Not Completed | 42

BASELINE CHARACTERISTICS:
Arm/Group | Vinflunine
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 18
Age Continuous [Mean (Standard Deviation); unit: years] | 61 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 28
Region of Enrollment [Number; unit: participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR), the Percentage of Patients Who Experience an Objective Benefit From Treatment
Description: Overall response rate is the percentage of patients with complete response or partial response per RECIST v.1 Criteria. Complete response (CR) = Disappearance of all target lesions, disappearance of all nontarget lesions for at least 4 weeks. Partial Response (PR) = At least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of longest diameters. The final response criteria assigned represented the best response obtained during treatment.
Time Frame: 18 months
Population: All patients were assessed for response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vinflunine
Number analyzed (Participants) | 51
percentage of participants | 19.6 [10 to 33]

2. Secondary Outcome: Duration of Response, the Length of Time, in Months, That Protocol Treatment Produced an Objective Improvement in Patients' Disease
Description: The Response Duration was calculated from time of initial measured response to date of first observation of progressive disease.
Time Frame: 18 months
Population: All patients were assessed for response. Only patients with objective response were analyzed for response duration.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vinflunine
Number analyzed (Participants) | 10
Months | 2.7 [1.9 to 3.9]

3. Secondary Outcome: Overall Survival (OS), the Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Death
Description: Overall survival was measured from the date of study entry until the date of death.
Time Frame: 18 months
Population: All patients were assessed for overall survival.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vinflunine
Number analyzed (Participants) | 51
Months | 4.9 [3.2 to 6.5]

4. Secondary Outcome: Progression Free Survival (PFS), the Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Worsening of Their Disease
Description: Progression free survival was defined as the interval between the start date of treatment and the date of occurrence of progressive disease or death.
Time Frame: 18 months
Population: All patients were assessed for progression free survival.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vinflunine
Number analyzed (Participants) | 51
Months | 1.6 [1.3 to 3.9]

ADVERSE EVENTS:
Arm/Group | Vinflunine
Serious Adverse Events (participants affected / at risk) | 31/51
Other Adverse Events (participants affected / at risk) | 30/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vinflunine (N=51)
Constipation (Gastrointestinal disorders) | 1 (1)
Death not associated with CTCAE term - Disease Progression NOS (General disorders) | 11 (11)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Failure to thrive (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Infection - Other (Pneumonia) (Infections and infestations) | 2 (2)
Altered Mental Status (Nervous system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)
Neutrophils (Blood and lymphatic system disorders) | 4 (4)
Obstruction, GI - Small Bowel NOS (Gastrointestinal disorders) | 1 (1)
Pain - abdomen (Gastrointestinal disorders) | 2 (2)
Pain - joint (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Other (Pain Syndrome) (General disorders) | 1 (1)
Pancreatic endocrine: glucose intolerance (Endocrine disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Supraventricular and nodal arrhythmia - Atrial Fibrillation (Cardiac disorders) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Leukocytes (Blood and lymphatic system disorders) | 2 (2)
Platelets (Blood and lymphatic system disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vinflunine (N=51)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (14)
Hemoglobin (Blood and lymphatic system disorders) | 28 (58)
Anorexia (Gastrointestinal disorders) | 16 (30)
AST (Metabolism and nutrition disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 30 (53)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (13)
Dehydration (Gastrointestinal disorders) | 5 (6)
Diarrhea (Gastrointestinal disorders) | 12 (15)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 19 (31)
Edema (Blood and lymphatic system disorders) | 3 (3)
Fatigue (General disorders) | 30 (71)
Fever (General disorders) | 7 (8)
Hyperglycemia (Metabolism and nutrition disorders) | 10 (25)
Hypertension (Cardiac disorders) | 3 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (8)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 4 (8)
Hyponatremia (Metabolism and nutrition disorders) | 8 (15)
Insomnia (General disorders) | 4 (8)
Leukopenia (Blood and lymphatic system disorders) | 15 (30)
Mucositis (Gastrointestinal disorders) | 4 (11)
Nausea (Gastrointestinal disorders) | 24 (39)
Nausea (intermittent) (Gastrointestinal disorders) | 4 (7)
Neuropathy (sensory) (Nervous system disorders) | 3 (4)
Neutropenia (Blood and lymphatic system disorders) | 21 (47)
Pain (General disorders) | 3 (5)
Pain (abdominal) (Gastrointestinal disorders) | 6 (6)
Pain (bone) (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain (chest) (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Pain (headache) (Nervous system disorders) | 3 (5)
Pain (jaw) (Musculoskeletal and connective tissue disorders) | 4 (4)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (21)
Vomiting (Gastrointestinal disorders) | 16 (23)
Vomiting (intermittent) (Gastrointestinal disorders) | 3 (5)
Weakness (General disorders) | 10 (17)
Weight Loss (General disorders) | 7 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.